CLINICAL TRIAL: NCT05696639
Title: Cerebral Venous Assessment on Brain Swelling in Patients With Aneurysm Subarachnoid Hemorrhage: Retrospective Cohort Study
Brief Title: SMCV Assessment on Brain Swelling in Patients With SAH
Acronym: Bayysmcv
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shenzhen Baoan District People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BYL20220216
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Aneurysm; Subarachnoid Hemorrhage; Brain Swelling
MeSH Terms: conditions — Aneurysm; Subarachnoid Hemorrhage; Brain Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Undeveloped venous group: patients with undeveloped cerebral venous
  Interventions: Procedure: Aneurysm embolization
- Well Developed venous group: patients with well-developed cerebral venous
  Interventions: Procedure: Aneurysm embolization

INTERVENTIONS:
Procedure: Aneurysm embolization — All patients underwent Aneurysm embolization surgery, the cerebral venous will be observed intraoperatively.

SUMMARY:
Cerebral swelling is a major complication following aneurysmal subarachnoid hemorrhage.This study is a retrospective cohort aimed to predict the extent of brain swelling. Cerebral venous assessment can identify the risk of brain swelling and improve surgical outcomes.

DETAILED DESCRIPTION:
Cerebral swelling is a major complication following aneurysmal subarachnoid hemorrhage (SAH).This study is a retrospective cohort aimed to predict the extent of brain swelling (BS). Cerebral venous assessment can identify the risk of cerebral swelling and improve surgical outcomes. This study is a retrospective cohort analysis. Cerebral venous angiography (CVA) will be adopted and the superficial middle cerebral vein (SMCVs) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

patients with anterior communicating aneurysm

Exclusion Criteria:

Hunt-Hess grade I- patients with posterior communicating aneurysm, poor general condition or combined with pregnancy , malignant tumors were excluded.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with an anterior communicating aneurysmal subarachnoid hemorrhage between January 2017 and December 2022 who underwent aneurysm embolization surgery, excluding patients with posterior communicating aneurysm, poor general condition or combined with pregnancy , malignant tumors.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
brain swelling | 2 weeks
  grading of brain swelling

CONTACTS AND LOCATIONS:
Overall Officials: JIangang Hu, Phd, Study Director — The People Hospital of Shenzhen Baoan
Locations (1):
- Shenzhen Baoan People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Y, Hu J. Effects of low-dose intravenous heparin therapy in aneurysmal subarachnoid hemorrhage: a randomized controlled clinical trial protocol. Trials. 2023 Jul 8;24(1):447. doi: 10.1186/s13063-023-07493-9. PMID 37422666